CLINICAL TRIAL: NCT02860429
Title: Clinical Trial of Cinobufacini Injection Combined With Oxaliplatin Regimen on Gastrointestine Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiaonan Cui (Other)
Responsible Party: Sponsor-Investigator, Xiaonan Cui, Professor,Chief Physician, The First Affiliated Hospital of Dalian Medical University
Organization: The First Affiliated Hospital of Dalian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCKY2016-37
Record Dates: First submitted 2016-08-01; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Gastrointestinal Neoplasms
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — huachansu; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cinobufacini injection (Experimental): Capsule Dosage and frequency:This group receives cinobufacini injection 20ml mixed with 5% Glucose injection 500ml started at the first day of chemotherapy until seven days once a day.
  Duration:6 chemotherapy cycles.
  Interventions: Drug: Cinobufacini injection; Drug: chemotherapy
- Control group (Other): Only receive the same chemotherapy with the experimental groups.No Cinobufacini injection.And have the same adjuvant treatment with the experimental groups.
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Drug: Cinobufacini injection — cinobufacini injection 20ml mixed with 5% Glucose injection 500ml started at the first day of chemotherapy until seven days once a day.
  Arms: Cinobufacini injection
Drug: chemotherapy — Chemotherapy is the oxaliplatin combination with fluorouracil regimen.

SUMMARY:
The clinical trail of Cinobufacini injection combined with Oxaliplatin regimen on gastrointestine carcinoma.This trail is randomized controled.Patients are diagnosed gastrointestinal cancer based on pathology or cell biology.They are randomized into 2 groups:both groups receive Oxaliplatin regimen.The treatment group receives Cinobufotalin 20ml mixed with 5% Glucose injection 500ml from the first day of chemotherapy until seven days in addition to the chemotherapy.The control group only receive the same chemotherapy with the treatment group.Both group have the same adjuvant therapy.Mainly to study of oxaliplatin into Cinobufacini injection leads to the influence of the peripheral nerve toxicity.Clinical evaluation includes neural electrophysiological test,chemotherapy drug toxicities,quality of life(QOL),etc.Blood biochemistry tests mainly include inflammatory cytokines,peroxidase reaction,immune cell number ratio and stress hormone,etc.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-70
* male and female
* signed the informed consent form.
* Diagnosis:Gastrointestinal cancer diagnosed by imaging,cell and pathology report.
* Eastern Cooperative oncology Group(ECOG)O-2,life expectancy more than 3 months.
* Indication for Chemotherapy,no contraindication.
* First time chemotherapy or at least 6 months after last chemotherapy and radiotherapy.
* At least 8 weeks after last biotherapy.
* Surgery:had not received transplantation surgery,at least 2 weeks after last major surgery.

Exclusion Criteria:

* Chemotherapy is contraindicated.
* Have the primary disease can cause the neuropathy.
* A history of other malignant tumor in recent 5 years.
* Less than 6 months after last chemotherapy or radiotherapy.
* Less than 8 weeks after last biotherapy.
* Cinobufotalin allergy.
* Had received transplantation surgery,less than 2 weeks after last major surgery.
* Other researchers think is not suitable for this clinical trail.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
neural electrophysiological test | every cycle of chemotherapy(measure 6 cycles,each cycle is 21days),up to 6 months

SECONDARY OUTCOMES:
The quality of life questionnaire(QLQ)-C30 | every cycle of chemotherapy(measure 6 cycles,each cycle is 21days),anticipate up to 5 months
National Cancer Institute(NCI)Common Toxicity Criteria | every cycle of chemotherapy(measure 6 cycles,each cycle is 21days),anticipate up to 5 months
Levi sensory nerve toxicity classification standard | every cycle of chemotherapy(measure 6 cycles,each cycle is 21days),anticipate up to 5 months
image test | For adjuvant chemotherapy patients every 3 months.For saving chemotherapy patients every 2 months.anticipate up to 1 years.
inflammatory cytokines,in blood. | every cycle of chemotherapy(measure 6 cycles,each cycle is 21days),anticipate up to 5 months
  For example:Interleukin(IL)-6,tumor necrosis factor(TNF)etc,in bood
peroxidase reaction,in blood. | every cycle of chemotherapy(measure 6 cycles,each cycle is 21days),anticipate up to 5 months
immune cell number ratio,in blood. | every cycle of chemotherapy(measure 6 cycles,each cycle is 21days),anticipate up to 5 months
stress hormone,in blood. | every cycle of chemotherapy(measure 6 cycles,each cycle is 21days),anticipate up to 5 months
  Estradiol(Female),testosterone(male)etc,in bood.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonan Cui, MD,PhD, Principal Investigator — The First Affiliated Hospital of Dalian Medical University; Rui Zhang, Principal Investigator — Liaoning cancer province
Locations (2):
- China (2):
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: Undecided